CLINICAL TRIAL: NCT01539473
Title: A Phase 1, Blinded, Placebo-Controlled, Crossover TR-701 FA Study of Blood Pressure Response Post-Tyramine Challenge
Brief Title: A Phase 1 TR-701 FA Study of Blood Pressure Response Post Tyramine Challenge
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: 1986-032; TR701-105 (Other: TriusRX Unique ID)
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Tyramine; tedizolid phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TR-701 FA with Tyramine (Experimental): TR-701 FA 200 oral with Tyramine
  Interventions: Drug: TR-701 FA with Tyramine
- Placebo-controlled with Tyramine (Placebo Comparator): Placebo-controlled with Tyramine
  Interventions: Drug: Placebo-controlled withTyramine

INTERVENTIONS:
Drug: TR-701 FA with Tyramine — TR-701 FA 200 mg oral and Tyramine
  Other Names: Tedizolid Phosphate
  Arms: TR-701 FA with Tyramine
Drug: Placebo-controlled withTyramine — Placebo-controlled and Tyramine
  Arms: Placebo-controlled with Tyramine

SUMMARY:
Phase 1 study to determine the effect of oral TR-701 FA on SBP response when administered with tyramine

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, 2-way crossover study to determine the effect of 200 mg oral TR-701 FA on SBP response when administered with tyramine in healthy adult male and female volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 to 45 years of age, inclusive
* Body mass index between 19 kg/m2 and 31 kg/m2, inclusive
* Healthy subjects with no clinically significant abnormalities identified by a detailed medical history,

Exclusion Criteria:

* Systolic blood pressure >130 mmHg or <90 mmHg measured after 10 minutes in the supine position at Screening or at admission to the study center
* Heart rate >90 bpm or <45 bpm measured after 10 minutes in the supine position
* Electrocardiogram (ECG) finding of QTc interval >500 msec, or other clinically significant ECG abnormality at the Screening Visit

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 14 days
  To assess tyramine dose required to cause increase of 30 mmHg in systolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Philippe G Prokocimer, MD, Study Chair — Trius Therapeutics
Locations (1):
- Trius Investigator Site 001, Evansville, Indiana, United States

REFERENCES:
- [Derived] Flanagan S, Bartizal K, Minassian SL, Fang E, Prokocimer P. In vitro, in vivo, and clinical studies of tedizolid to assess the potential for peripheral or central monoamine oxidase interactions. Antimicrob Agents Chemother. 2013 Jul;57(7):3060-6. doi: 10.1128/AAC.00431-13. Epub 2013 Apr 22. PMID 23612197